CLINICAL TRIAL: NCT07203664
Title: Use of Tacrolimus and MTOR Inhibitors With Anticipatory Therapy vs. Tacrolimus and Mycophenolic Acid With Universal Prophylaxis in Renal Recipients at High Risk of Posttransplant Cytomegalovirus. Phase 4 Clinical Trial. TIMTOR STUDY.
Brief Title: Use of Tacrolimus and MTOR Inhibitors With Anticipatory Therapy vs. Tacrolimus and Mycophenolic Acid With Universal Prophylaxis in Renal Recipients at High Risk of Posttransplant Cytomegalovirus.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, María Ovidia López Oliva, Dra., Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TIMTOR
Record Dates: First submitted 2025-09-09; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Evaluate the Effectiveness of CMV Prevention Strategies in Kidney Transplant Recipients
MeSH Terms: interventions — Steroids; Tacrolimus; MTOR Inhibitors; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: exploratory, randomised, open-label, single-centre trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mTOR inhibitors (Experimental): Preemptive therapy will be administered as a preventive strategy, consisting of initiating antiviral treatment with valganciclovir (900 mg every 12 hours, adjusted according to renal function as per the technical data sheet) when CMV viral replication in blood exceeds 1,000 copies/ml. Treatment will be discontinued once viral load becomes undetectable in two consecutive tests
  Interventions: Combination Product: steroids, tacrolimus and mTOR inhibitors
- Universal prophylaxis (Active Comparator): As a preventive strategy against CMV, the patient will receive universal prophylaxis, and for maintenance immunosuppressive treatment, steroids, tacrolimus, and mycophenolic acid will be administered.
  Interventions: Combination Product: steroids, tacrolimus and mycophenolic acid.

INTERVENTIONS:
Combination Product: steroids, tacrolimus and mTOR inhibitors — Patients receive immunosuppressive induction treatment with thymoglobulin (at least 1 dose and maximum of 5 doses) and immunosuppressive maintenance treatment with tacrolimus + mTOR inhibitors. Preemptive therapy will be administered as a preventive strategy, consisting of initiating antiviral treatment with valganciclovir (900 mg every 12 hours, adjusted according to renal function as per the technical data sheet) when CMV viral replication in blood exceeds 1,000 copies/ml. Treatment will be discontinued once viral load becomes undetectable in two consecutive tests.
  Arms: mTOR inhibitors
Combination Product: steroids, tacrolimus and mycophenolic acid. — Patients will receive immunosuppressive induction treatment with thymoglobulin (at least 1 dose and a maximum of 5 doses) and tacrolimus + mycophenolic acid following the guidelines of the technical file and the centre's usual protocols.
  Arms: Universal prophylaxis

SUMMARY:
The overall objective of this project is to optimise preventive treatment of CMV infection/disease in renal transplant recipients at increased risk of CMV post-transplantation. The specific objectives are: (1) To compare the incidence of CMV infection/disease at 6 months post-transplant in Ig G CMV positive (R+CMV) recipients receiving induction treatment with thymoglobulin and one of the two maintenance immunosuppressive treatment regimens used in routine clinical practice : tacrolimus and MTOR inhibitors (group 1) or tacrolimus and mycophenolic acid (group 2); (2) To monitor CMV-specific cellular immunity before transplantation, at 15, 30 and 90 days post-transplantation. For this purpose, an exploratory phase 4 clinical trial has been designed in which will select 30 R+CMV patients receiving renal transplantation with induction treatment with thymoglobulin. After signing informed consent, patients will be randomised to receive one of the two immunosuppression regimens indicated above. The patients in group 1 will receive early therapy as a CMV prevention strategy and patients in group 2 will receive universal prophylaxis for 3 months. Follow-up visits to will be conducted according to the usual protocol and clinical and virological variables will be collected. In addition, blood samples will be collected for the assessment of CMV-specific cellular immunity before and after transplantation. The primary endpoint is the presence of CMV infection/disease post-renal transplantation at 6 months. Secondary variables include renal function, acute rejection, patient and graft survival and the occurrence of surgical or haematological complications.

DETAILED DESCRIPTION:
HYPOTHESIS The use of immunosuppressive maintenance therapy including mTOR inhibitors versus the use of mycophenolic acid in kidney transplant patients with an increased risk of post-transplant CMV disease (R+CMV receiving induction with thymoglobulin) will allow optimisation of the preventive treatment of these patients, presenting a similar incidence of post-transplant CMV disease in both groups and better maintenance of CMV-specific cellular immunity post-transplant.

OBJECTIVES General Objective: To improve the preventive treatment of CMV disease in renal transplant patients at increased risk.

Main Objectives: (1) To compare the incidence of CMV disease at 6 months post-renal transplant in Ig G CMV-positive recipients receiving induction treatment with thymoglobulin and maintenance treatment with tacrolimus and mTOR inhibitors (group 1) with CMV prevention strategy of anticipatory therapy or tacrolimus and mycophenolic acid (group 2) with CMV prevention strategy with universal prophylaxis. (2) Monitor CMV-specific cellular immune response before transplantation and at 15, 30 and 90 days post-transplantation in each of the two treatment groups using Quantiferon-CMV.

Secondary Objectives: (3) To compare between the two groups the incidence of CMV infection, delayed initial graft function, acute rejection diagnosed by renal biopsy, renal function and patient and graft survival in the first 6 months post-transplant. (4) To compare between the two groups the presence of surgical (lymphocele requiring intervention) or haematological (neutropenia) complications in the first 6 months post-transplantation.

STUDY DESIGN Phase IV, exploratory, randomised, open-label, single-centre, exploratory clinical trial to evaluate the effectiveness of CMV prevention strategies comparing early therapy vs. universal prophylaxis in Ig G CMV-positive kidney transplant recipients treated with thymoglobulin receiving tacrolimus and mTOR inhibitors (group 1) vs. tacrolimus and mycophenolic acid (group 2).

Patients who meet the inclusion criteria and who sign the informed consent form the day before transplant surgery (pre-transplant day) will have a blood sample taken for CMV-specific cellular immunity analysis using quantiferon CMV and will be randomised into two groups on the day of renal transplant surgery (day 0).

a) Group 1: Will receive, as a CMV prevention strategy, early therapy, and as maintenance immunosuppressive treatment steroids, tacrolimus and mTOR inhibitors. b) Group 2: Will receive, as a CMV prevention strategy, universal prophylaxis, and as maintenance immunosuppressive therapy steroids, tacrolimus and mycophenolic acid. A randomisation list will be generated using SAS 9.4. software, in order to achieve a balanced randomisation in the treatment groups. The ratio will be 1:1 for each group and stratified by sex.

Definition of the groups: Group 1: Will receive early therapy, as a prevention strategy, which consists of starting antiviral treatment with valganciclovir (900 mg/12 hours, adjusted to renal function, according to the technical data sheet) when CMV viral replication is detected in blood above 1,000 copies/ml and treatment will be suspended when the viral load is negative in two consecutive controls.

Group 2: will receive universal prophylaxis with valganciclovir (900 mg/24 hours, adjusted to renal function, according to technical data sheet) during the first 3 months post-transplant, as a CMV prevention strategy.

All patients will receive immunosuppressive induction treatment with thymoglobulin (at least 1 dose and a maximum of 5 doses) and immunosuppressive maintenance treatment with tacrolimus + mTOR inhibitors (patients in group 1) or tacrolimus + mycophenolic acid (patients in group 2) following the guidelines of the technical file and the centre's usual protocols.

Follow-up visits will be performed at 15, 30, 90, 120, 120, 150 and 180 days post-transplant where clinical, analytical, virological (CMV viral loads by PCR in whole blood) and immunological (analysis of CMV-specific cellular immunity by CMV quantiferon) data of the patients will be evaluated. Data on the presence or absence of CMV infection or disease at each visit, concomitant medication changes and adverse events will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more.
* Positive pre-transplant Ig G CMV serology.
* Receive immunosuppressive induction treatment with thymoglobulin (between 1 and 5 doses).
* Agree to participate in the study by signing the informed consent form.

Exclusion Criteria:

* Patients with negative pre-transplant Ig G CMV serology.
* HIV-infected patients.
* Patients receiving induction therapy with basiliximab.
* Patients who cannot comply with the follow-up protocol.
* Patients who cannot receive iMTOR as initial maintenance immunosuppressive therapy, such as patients with chronic kidney disease secondary to hepatorenal polycystic kidney disease and patients who are expected to undergo complex vascular surgery.
* Patients who for any reason should not be included in the study according to the evaluation of the research team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CMV disease incidence | 6 months after renal transplant
  To compare the incidence of CMV disease at 6 months post-renal transplantation in Ig G CMV-positive recipients receiving induction treatment with thymoglobulin and maintenance treatment with tacrolimus and mTOR inhibitors (group 1) with CMV prevention strategy of early therapy or tacrolimus and mycophenolic acid (group 2) with CMV prevention strategy with universal prophylaxis.
Monitor CMV-specific cellular immune response prior to transplantation | 4 months
  Monitor CMV-specific cell-mediated immune response before transplantation and at 15, 30 and 90 days post-transplantation in each of the two treatment groups using Quantiferon-CMV.

SECONDARY OUTCOMES:
To compare between the two groups the incidence of CMV infection, delayed initial graft function, acute rejection diagnosed by renal biopsy, renal function and patient and graft survival | 6 months
  To compare between the two groups the incidence of CMV infection, delayed initial graft function, acute rejection diagnosed by renal biopsy, renal function and patient and graft survival in the first 6 months post-transplantation.
To compare the presence of surgical (lymphocele requiring intervention) or haematological (neutropenia) complications | 6 months
  To compare between the two groups the presence of surgical (lymphocele requiring intervention) or haematological (neutropenia) complications in the first 6 months post-transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Pº de la Castellana, 261 (Servicio de Nefrologia), Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No